CLINICAL TRIAL: NCT07191145
Title: EarLy Infusion of Eptinezumab for TreatmEnt of ACute Post-Traumatic Headaches (ELITE-ACT): a Parallel Group, Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Eary Infusion of Eptinezumab for TreatmEnt of ACute Post-Traumatic Headaches (ELITE-ACT)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6558
Record Dates: First submitted 2025-09-05; First posted 2025-09-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Headache
Keywords: Migraine
MeSH Terms: conditions — Post-Traumatic Headache; Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Intervention Model Description: Group 1: Intervention - Eptinzumab 300mg IV once within 8 weeks of PTH onset Group 2: Control - Placebo once within 8 weeks of PTH onset
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Eptinezumab (Experimental): Eptinezumab 300mg IV once within 8 weeks of post-traumatic headache onset
  Interventions: Drug: Eptinezumab
- Control - Placebo (Placebo Comparator): Placebo IV once within 8 weeks of post-traumatic headache onset
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab 300mg IV
  Arms: Intervention - Eptinezumab
Other: Placebo — Control - placebo IV
  Arms: Control - Placebo

SUMMARY:
Most individuals with mild traumatic brain injury (mTBI) experience post-traumatic headaches (PTH). Of PTH, 50% present with a migraine phenotype which is the most disabling type of PTH. Patients with migraine-PTH are at greater risk of persistent symptoms whereby the acute PTH (aPTH) becomes persistent PTH (pPTH) (ie. lasting > 3 months) with a conversion rate of 47-95%. As migraine symptoms become chronic, it becomes treatment resistant. Despite these implications, early preventive medication management of PTH is marred by lengthy trials of multiple medications (2-3 months for each) and adverse effects that aggravate mTBI symptoms (fatigue, nausea, and presyncope). There is a compelling need to establish an effective treatment to prevent this debilitating outcome. Eptinezumab is a calcitonin gene-related peptide (CGRP)-blocking monoclonal antibody that reduces migraine burden in patients with migraines after a single infusion. Patients with PTH have higher serum levels of CGRP and experimental infusion of CGRP to patients with mTBI reproduces migraine PTH symptoms. Given the similarly in CGRP expression between chronic migraines and PTH, an infusion of eptinezumab within 8 weeks of PTH is hypothesized to reduce headache burden 3 months after treatment and prevent pPTH.

DETAILED DESCRIPTION:
Approximately 500,000 Canadians aged >12 experienced a mild traumatic brain injury (mTBI) in the preceding year based on a 2020 report. Patients with mTBIs have a cumulative incidence of headaches, termed post-traumatic headaches (PTH), of 91% over one year following injury. Post-traumatic headache (PTH), according to the International Classification of Headache Disorders (ICHD) by definition, is a headache caused by a traumatic injury to the head. This condition is further classified into acute PTH (aPTH) which is a headache of less than 3 months duration following injury to the head, and persistent PTH (pPTH) which refers to the transition of aPTH to longer than 3 months duration.

PTH is the most common symptom after mTBI. The impact of PTH is significant as the majority of patients with aPTH (up to 95%) transition to pPTH. In patients who experience PTH, the frequency of headache burden may vary with one study reporting a mean monthly headache frequency of 25 days. Individuals with PTH have decreased cognitive function with impaired memory tests, slower reaction, and struggle in returning to their previous physical and social functions. Therefore, PTH has a profound emotional, social, and economic impact. Treatment for PTH is currently guided by its phenotype - migraine, tension, or trigeminal autonomic cephalgias. PTH with migraine phenotype occurs in 49% of cases and tension phenotype in 40%, whereas 11% are undefined. Patients with tension-PTH are by definition headaches with mild to moderate intensity, whereas patients with migraine-PTH are categorized as severe. Patients with migraine-PTH are more likely to have near daily headaches and have a higher probability of progressing to pPTH.

The pathophysiology of migraine-PTH results from activation of the trigeminovascular system (TVS). Release of CGRP from the TVS has been identified as the primary mechanism where increased sensitivity of trigeminal nociceptors that innervate the dura mater is responsible for intracranial pain. As migraine progresses, frequent and sustained activation of the TVS and its central connections may lead to neuroplastic changes and a reduced threshold for initiating migraine attacks. Patients with PTH are known to have higher serum levels of CGRP and infusion of CGRP to patients with mTBI reproduces migraine PTH symptoms. Current evidence on treatment of PTH is limited to two placebo-controlled trials involving botulinum toxin and fremanezumab. Both trials involved patients that had established and pPTH and neither specifically selected for patients with migraine-PTH to the best of our knowledge (fremanezumab study is unpublished). The fremanezumab study also did not demonstrate a significant improvement compared to placebo in the pPTH population. A third open label study on pPTH and erenumab demonstrated a reduction of 2.8 days per month in a 12 week trial and was well-tolerated.

There is pre-clinical evidence demonstrating early administration of CGRP-blocking monoclonal antibodies (MAb) is important to prevent establishment of central sensitization after mTBI. Once central sensitization is established, additional CGRP-independent mechanisms promote or maintain central sensitization and CGRP-blocking MAbs are less effective. Therefore, there has been a focus to target aPTH prior to progression to pPTH. The American Headache Society's recent position statement endorsed the use of CGRP-targeting therapies, including MAbs, as first-line options due to their efficacy across multiple patient-important outcomes and favourable safety profile. CGRP-targeting therapies have excellent tolerability and efficacy evidenced by low drop out rates. There are currently two trials registered on www.ClinicalTrials.gov assessing erenumab, a subcutaneously administered CGRP-blocking monoclonal antibody, for treatment of aPTH that are in progress. Notably, both trials have pursued all phenotypes of PTH rather than migraine-PTH to which CGRP MAb is specific for treating.

Eptinezumab is a CGRP-blocking MAb approved by Health Canada for prevention of migraines in patients with greater than 4 migraine days per month. It is unique as the only intravenously administered CGRP MAb. It has superior bioavailability (100% after 30 min infusion achieving maximum plasma concentration with the first dose) and as a single dose, versus monthly subcutaneous injection of erenumab, has higher medication compliance. The Health Canada recommended doses are 100mg or 300mg. Large scale randomized controlled trials have been conducted comparing eptinezumab to placebo in patients with episodic and chronic migraine. These trials showed that monthly migraine days (MMD) were reduced 0.7 to 2.7 days at 12 weeks for the 100 mg dose and 1.0 to 3.2 days for the 300 mg dose compared to placebo. Eptinezumab has been shown to have greater proportions of reductions of 50% in MMD in the first 12 weeks compared to placebo and also a greater proportion of patients who experienced 100% reduction in MMD at 12 weeks than placebo. A recent meta-analysis demonstrated that compared to eptinezumab 100mg, the 300mg dose was associated with substantially reduced MMD with no significant differences in adverse events or serious adverse events.

The most common adverse effects reported with eptinezumab use included upper respiratory tract infections, hypersensitivity or infusion site reactions, nasopharyngitis, nausea, and sinusitis. In post-marketing surveillance, 10.4% of patients reported mild adverse effects including vertigo, constipation, rhinitis, myalgia, weight gain, hoarseness, and hypotension. Hypersensitivity reactions include angioedema, urticaria, flushing, rash, and pruritus (reported in 3-4% of patients). The only absolute contraindication to eptinezumab is hypersensitivity to the active substance or any of the excipients. Eptinezumab contains sorbitol and therefore patients with Hereditary Fructose Intolerance should not receive it.

In the PTH population where memory impairment can be an issue, eptinezumab has the added benefit of prolonged duration of therapeutic benefit (3 vs 1 month compared to other subcutaneous injectable CGRP MAbs) thereby resulting in decreased dosing frequency and increased compliance. Eptinezumab also has the added advantage of rapid onset which has been observed on day 1 post-treatment whereas other MAbs may take 1 month or more to establish benefit. The rapid onset of effect may prove to be advantageous to prevent progress from aPTH to pPTH. Given its ease of use as a rapid-acting single-administration medication, evidence in reduction in MMD, good tolerability and safety profiles, and adherence to treatment (single IV versus multiple doses), eptinezumab is an ideal candidate for study in patients with migraine-PTH.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for acute post-traumatic headache as per ICHD-3 criteria
* Meet migraine screening questionnaire criteria (MSQ score ≥ 4) during at least one of the weekly screening calls
* Within 8 weeks after onset of PTH

  * Imaging is not required for inclusion
* Negative human chorionic gonadotropin test before treatment, for female participants of childbearing potential who are not practicing medically appropriate methods of birth control (e.g., hormonal contraceptives, implants, injectables, intrauterine devices, intrauterine systems, etc.)

Exclusion Criteria:

* Diagnosis of moderate to severe TBI
* History of mTBI within the past 5 years
* Pre-existing chronic migraine and its subtypes, tension-type headache, trigeminal autonomic cephalalgias, cranial neuralgias, daily headache, diagnosis of another secondary headache disorder per ICHD-3 (except medication overuse headache)
* Concurrent use of CGRP-related treatment or botulinum toxin within the last three month for migraine
* Substance / opioids use disorder
* Confounding chronic pain disorder / clinically significant pains
* Concurrent major injuries (long bone, rib, and spinal fractures) or surgical intervention while in hospital on initial trauma
* On-going litigation for current trauma
* Pregnancy/breast-feeding
* Uncontrolled psychiatric conditions (depression, PTSD, anxiety, functional neurological disorder)
* Use of opioids/barbiturates for headaches (> 4 days/month)
* Hereditary fructose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Headache frequency | 9-12 weeks (inclusive) after intervention
  Number of moderate to severe headache days between 9-12 weeks (inclusive) after intervention

SECONDARY OUTCOMES:
Responder rate | At 9-12 weeks (inclusive) after treatment, those reporting a 50% reduction from baseline are considered responders.
  Percentage change from baseline in the number of moderate to severe headache days, as captured by the participant's headache diary and at weekly follow-ups. At 9-12 weeks (inclusive) after treatment, those reporting a 50% reduction from baseline are considered responders.
Acute treatment utilization | Daily until 12 weeks
  The number of days in which an acute headache treatment was used, as captured daily in the participant headache diary, at baseline, and at weekly follow-ups until week 12.
Preventive treatment utilization | Daily until 12 weeks
  The utilization of preventive analgesics, as a categorical yes/no variable, will be recorded daily in the participant headache diary, at baseline and at weekly follow-ups until week 12
Headache disability | Baseline until 12 weeks
  Patient-reported disability due to their headache, assessed using the Headache Impact Test (HIT-6) at baseline and during follow-ups at 4/8/12/24 weeks. Minimum score 36, maximum score 78; higher score indicates worse outcome.
Concussion severity | Baseline until 12 weeks
  Patient-reported disability due to their headache, assessed using the Rivermead Post-Concussion Symptoms Questionnaire (RPQ), at baseline and during follow-ups at 4/8/12 weeks. Minimum score 0, maximum score 52; higher score indicates worse outcome.
Emotional Function | Baseline until 12 weeks
  Patient-reported anxiety using General Anxiety Disorder scale (GAD-7) at baseline and during follow-ups at 4/8/12 weeks. Minimum score 0, maximum score 21; higher score indicates worse outcome.
Emotional Function | Baseline until 12 weeks
  Patient-reported mood using the Patient Health Questionnaire (PHQ-9) at baseline and during follow-ups at 4/8/12 weeks. Minimum score 0, maximum score 27; higher score indicates worse outcome.
Emotional Function | Baseline until 12 weeks
  Patient-reported post-traumatic stress using the PTSD checklist for DSM-5 (PCL-5) at baseline and during follow-ups at 4/8/12 weeks. Minimum score 0, maximum score 80; higher score indicates worse outcome.
Patient satisfaction | Baseline until 12 weeks
  Patient-reported satisfaction with their treatment, assessed using the patient global impression of change (PGIC), at baseline and during follow-ups at 4/8/12 weeks. Minimum score 0, maximum score 10; higher score indicates worse outcome.
Sleep quality | Baseline until 12 weeks
  Patient-reported sleep quality, assessed using the PROMIS 6a sleep questionnaire at baseline and during follow-ups at 4/8/12 weeks. Minimum score 6, maximum score 30; higher score indicates worse outcome.

OTHER OUTCOMES:
Adverse events | Baseline until until 24 weeks after treatment
  Adverse events related to study medication

CONTACTS AND LOCATIONS:
Overall Officials: Howard Meng, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication, no limit on time
Access Criteria: Contact study investigators